# **Statistical Analysis Plan**





# **TREATT**

# Trial to EvaluaAte Tranexamic acid therapy in Thrombocytopenia

Version: Final 1.1

Date: 13/03/2020

CTU Ref: 12-01-CSU ISRCTN: 73545489 REC: 14/SC/1290

MHRA CTA: 25224/0002/001-0001

Prepared by:

| Name | Role | Signature | Date |
|---------------|--------------------|-----------|------------|
| Elinor Curnow | Trial Statistician | | 13/03/2020 |

Approved by:

| Name | Role | Signature | Date |
|-----------------|--------------------|-------------------------|------------|
| Simon Stanworth | Chief Investigator | Approved electronically | 13/05/2020 |
| Lise Estcourt | Chief Investigator | Approved electronically | 13/05/2020 |
| lan Franklin | TSC Chair | Approved electronically | 02/07/2020 |
| Helen Thomas | Lead Statistician | Approved electronically | 17/06/2020 |

# **Statistical Analysis Plan**

# **Table of Contents**

| 1 | Background and Design | page 3 |
|---|--------------------------------------|---------|
| 2 | Outcome Measures | page 7 |
| 3 | Data Handling | page 8 |
| 4 | Detailed Analysis Plan | page 12 |
| 5 | Data Analysis Tables to be Completed | page 19 |
| 6 | Statistical Analysis Plan Amendments | page 36 |
| 7 | References | page 37 |

# **Statistical Analysis Plan**

#### 1. Background and Design

The main characteristics of this trial have been summarised using the TREATT Protocol v3.1 from 09/08/2018. Please refer to this Protocol for full details. All essential documents for the trial are held in the Trial Master File.

### 1.1 Trial Summary and Objective

# Background

Platelet transfusions are commonly administered as prophylaxis to reduce the risk of bleeding in patients with haematological malignancies. Two recent randomised controlled trials of prophylactic platelet transfusions have directly evaluated the benefit of prophylactic platelet transfusions more directly; both found a no-prophylaxis approach led to greater rates of World Health Organization (WHO) grade 2-4 bleeding overall. However although patients who received prophylactic platelet transfusions had fewer bleeds, a high baseline bleeding rate remained (43% of patients had WHO grade 2-4 bleeding in TOPPS¹). This suggests that factors other than those addressed by the use of platelet transfusions are important in determining bleeding risk.

A recent systematic review of clinical trials of tranexamic acid (TXA) in patients with haematological disorders to prevent bleeding identified 4 trials (published in 5 papers). All studies were small and of poor quality; all but one of the trials were conducted and published well over 10 years ago. The results suggest a reduction in bleeding, but it was not possible to combine the data. All studies reported a reduction in platelet usage. The trials were too small to assess the effect of TXA on thromboembolic events. For all these reasons, we believe that the effectiveness and safety of TXA in haematology is uncertain and that a high quality randomised controlled trial is needed.

#### Aim of study

To assess whether TXA reduces bleeding in haematology patients. Secondary outcomes include safety (thrombotic events) and platelet use.

#### 1.2 Patient Eligibility Criteria

#### Patient inclusion criteria:

Patients are eligible for this trial if:

- Aged ≥ 18 years of age
- Confirmed diagnosis of a haematological malignancy
- Undergoing, or planning to undergo, chemotherapy or haematopoietic stem cell transplantation
- Anticipated to have a hypoproliferative thrombocytopenia resulting in a platelet count of ≤ 10x10<sup>9</sup>/L for ≥ 5 days
- · Able to comply with treatment and monitoring

#### Patient exclusion criteria:

A patient will not be eligible for this study if he/she fulfils one or more of the following criteria:

1. Patients with a past history or current diagnosis of arterial or venous thromboembolic disease including myocardial infarction, peripheral vascular disease and retinal arterial or venous thrombosis.

# **Statistical Analysis Plan**

- 2. Diagnosis of acute promyelocytic leukaemia (APML) and undergoing induction chemotherapy
- 3. Patients with a diagnosis/previous history of veno-occlusive disease (also called sinusoidal obstruction syndrome)
- 4. Patients with known inherited or acquired prothrombotic disorders e.g.
  - a. Lupus anticoagulant
  - b. Positive antiphospholipids
- 5. Patients receiving any pro-coagulant agents (e.g. DDAVP, recombinant Factor VIIa or Prothrombin Complex Concentrates (PCC) within 48 hours of enrolment, or with known hypercoagulable state
- 6. Patients receiving L-asparaginase as part of their current cycle of treatment
- 7. History of immune thrombocytopenia (ITP), thrombotic thrombocytopenic purpura (TTP) or haemolytic uraemic syndrome (HUS)
- 8. Patients with overt DIC (See Appendix 3 in the protocol for definition)
- 9. Patients requiring a platelet transfusion threshold >10x10<sup>9</sup>/L at time of randomisation. (This refers to patients who require their platelet count to be maintained at a certain specified level on an ongoing basis, and excludes a transient rise in the threshold due to sepsis.)
- 10. Patients with a known inherited or acquired bleeding disorder e.g.
  - a. Acquired storage pool deficiency
  - b. Paraproteinaemia with platelet inhibition
- 11. Patients receiving anticoagulant therapy or anti-platelet therapy
- 12. Patients with visible haematuria at time of randomisation
- 13. Patients with anuria (defined as urine output < 10 mls/hr over 24 hours).
- 14. Patients with severe renal impairment (eGFR ≤30 ml/min/1.73m²)
- 15. Patients with a previous history of epilepsy, convulsions, fits or seizures
- 16. Patients who are pregnant or breast-feeding
- 17. Allergic to tranexamic acid.
- 18. Patients enrolled in other trials involving platelet transfusions, anti-fibrinolytics, platelet growth factors or other pro-coagulant agents.
- 19. Patients previously randomised into this trial at any stage of their treatment

# 1.3 Trial Intervention

#### Administration of Trial treatment

Trial treatment will be started as per randomisation assignment. Either as soon as possible within 24 hours, and no later than 72 hours, of the first recorded platelet count  $\leq 30 \times 10^9$ /L,

OR if the participant was admitted with a platelet count already below  $30 \times 10^9$ /L as soon as possible within 24 hours, and no later than 72 hours after the start of chemotherapy or conditioning for a stem cell transplant,

# All participants will start with Intravenous administration

The trial treatment (Tranexamic acid 1g /placebo) will be administered intravenously as a slow IV bolus over 10 minutes every 8 hours.

If the participant is well enough they can switch to:

#### Oral administration

The trial treatment (Tranexamic acid 1.5g/placebo) will be administered orally as a capsule/tablet every 8 hours.

TREATT\_SAP\_v1.1\_2020\_03\_13 Cross-Referenced in Primary Document: MPD998Page 4 of 38

# **Statistical Analysis Plan**

Figure 1 Summary of trial entry, randomisation and treatment



# **Statistical Analysis Plan**

#### 1.4 Randomisation and Blinding Procedures

Participants will be randomised to antifibrinolytic therapy or placebo in a 1:1 fashion, stratified by site. Randomisation will further be balanced within blocks of varying, undisclosed sizes. Randomisation lists will be created using computed-generated random numbers.

#### 1.5 Sample size calculation

### 1.5.1 Minimal Clinically Important Difference (MCID)

Based on the experience of similar patients in the TOPPS trial<sup>1</sup>, in the absence of antifibrinolytic therapy, it is anticipated that 43% of eligible patients would experience death or WHO Grade 2 bleeding or higher within the first 30 days. In such a background setting of bleeding, the trial investigators anticipate less than a 10% relative reduction in bleeding rates would not be sufficient to substantially change clinical practice, because the absolute risk reduction of 4.3% would mean that it would be necessary to treat approximately 23.3 patients in order for the treatment to have an impact on 1 patient ("Number Needed to Treat" (NNT) = 23.3).

As much as a 26% relative reduction in bleeding rates would likely be judged sufficient to change clinical practice, because the associated NNT = 8.9 patients might be acceptable, provided no new safety issues related to anti-fibrinolysis in the thrombocytopenic population are uncovered.

We thus evaluate the planned sample size of the trial relative to these hypothesised effects as a reference.

#### 1.5.2 Primary efficacy outcomes

616 participants will be accrued to the UK/Australian clinical trial.

The participants will be randomised in a double blind fashion to receive TXA or a matching placebo.

The clinical trial will be conducted with the primary endpoint of decreased proportion of death or WHO Grade 2 or higher bleeding among all participants receiving TXA versus placebo over 30 days. The type 1 error will be controlled at a two-sided level of 0.05. The primary endpoint will be analysed using the Kaplan-Meier (KM) method to estimate the probability of bleeding or death within 30 days in the analysis populations. Power and sample size calculations are based on a log-rank test for comparing two survival curves, as described in Collett<sup>2</sup>.

It is anticipated that the UK and Australia will be able to recruit 616 participants for this trial. Under the assumption that anti-fibrinolysis results in a decrease of death or WHO Grade 2 bleeding from 43% to 32%, the 616 participants will provide 80% power to detect an observed absolute decrease in bleeding rates of 11% (a relative reduction of 26% with a NNT of 8.9) and will be judged statistically significant at the two-sided 0.05 level. The planned trial size of 616 subjects includes an additional 5% of participants above the required sample size of 586. This 5% figure is more than the proportion of participants within TOPPS (4%) that dropped their platelet count below 50 x  $10^9$ /L but did not drop their platelet below 30 x  $10^9$ /L. This therefore accounts for the number of participants within the trial who are randomised but never receive the trial treatment.

We do not expect there to be a problem with the assessment of the primary outcome of bleeding over the 30 day trial period, starting from the first day of administration of the study intervention. In the recent TOPPS trial, completeness of bleeding outcome documentation was

# **Statistical Analysis Plan**

excellent. A bleeding assessment was completed on 93% (8405/9030) of days for participants in the no-prophylaxis group, and 97% (8733/8970) of days in the prophylaxis group. The majority of participants in both arms had bleeding information completed on each trial day (median no-prophylaxis 30 days (IQR 29 to 30); median prophylaxis 30 days (IQR 30 to 30)). There were also only 6 deaths (1% of participants) while on the trial.

#### 1.5.3 Safety outcomes

This trial is not powered to definitively establish the safety of the treatment with respect to the frequency of venous thromboembolism (VTE). However, with the planned enrolment of 616 participants, an observed difference in frequency of VTE of 3.6% on the placebo arm and 5% or less on the TXA arm would result in a 95% confidence interval that excluded a relative risk of 3.5.

#### 2. Outcome Measures

#### 2.1 Primary outcome measures

Estimated proportion of participants who died or had bleeding of WHO grade 2 or above during the first 30 days of the trial **from the first day of administration of the study intervention.** 

# 2.2 Secondary outcome measures

### 2.2.1 Secondary Efficacy Outcomes

All measured during first 30 days of the trial, i.e. from the first day of administration of the study intervention.

- Proportion of days with bleeding (WHO grade 2 or above)
- Time to first episode of bleeding of WHO grade 2 or greater for those participants who bled
- Highest grade of bleeding a participant experiences
- Number of platelet transfusions/participant
- Number of red cell transfusions/participant
- Proportion of participants surviving up to 30 days without a platelet transfusion
- Proportion of participants surviving up to 30 days without a red cell transfusion
- Quality of life

# 2.2.2 Secondary Safety Outcomes

- Number of thrombotic events from first administration of trial treatment up to and including
   120 days after the first dose of trial treatment is administered, per day at risk
- Number of participants developing Veno-occlusive Disease (VOD; Sinusoidal obstructive syndrome, SOS) within 60 days of first administration of trial treatment
- All-cause mortality during the first 30 days and the first 120 days after the first dose of trial treatment is administered
- Death due to thrombosis during the first 120 days after the first dose of trial treatment is administered
- Death due to bleeding during the first 30 days after the first dose of trial treatment is administered

# **Statistical Analysis Plan**

 Number of serious adverse events from first administration of trial treatment until 60 days after the first dose of trial treatment is administered

#### 2.2.3 Other Outcomes

All measured during first 30 days of the trial, i.e. from the first day of administration of the study intervention.

- Proportion of days with thrombocytopenia (≤10x10<sup>9</sup>/L, ≤30x10<sup>9</sup>/L, ≤50x10<sup>9</sup>/L)
- Proportion of days with fever (highest daily temperature ≥ 38.1°C) of days spent in hospital, up to study day 30
- · Reasons for platelet and red cell transfusions

#### 2.3 Sub-group analyses

Subgroup analyses will be performed for the primary outcome for the following variables in the main analysis:

- Country of participant (UK vs. Australia), if evidence of heterogeneity between UK and Australian participants is identified in the interim analysis
- Platelet count at consent (≤30x10<sup>9</sup>/L vs. > 30x10<sup>9</sup>/L)
- Treatment compliance during first 30 days of the trial (participant decided to stop taking trial treatment vs. participant did not decide to stop taking trial treatment)

### 3. Data Handling

3.1 CRF descriptions and data collection schedule

Table 1 CRF completion requirement

| CRF | Completion requirement |
|---|---|
| Form 1a- Eligibility & consent | Mandatory at consent |
| Form 2- Demography | Mandatory at consent |
| Form 3- Diagnosis & treatment plan | Mandatory at consent |
| Form 4- Medical history | Mandatory at consent |
| Form 5a- Laboratory data | Mandatory at consent |
| Form 5b- Laboratory data | Days between consent and randomisation |
| Form 6- Randomisation | Mandatory at randomisation |
| Form 7- Daily bleeding and Temperature assessment | From day R up to study day 30 |
| Form 8- Non-severe bleeding assessment | From day R up to study day 30, if non-<br>severe bleeding is reported on form 7b |

# **Statistical Analysis Plan**

| Form 9a- Severe bleeding assessment (initial report) | From day R up to study day 30, if severe bleeding is reported on form 7b |
|---|---|
| Form 9b- Severe bleeding assessment (follow-up report) | When form 9a has been completed |
| Form 10- Transfusion data form | From day R up to study day 30, if transfusion reported on form 6, form 7, form 12 or form 13 |
| Form 11- Interventions & procedures for daily bleeding | From day R up to study day 30, if indicated on form 7 |
| Form 12- Daily assessments | After day R, up to day 1 |
| Form 1b- Eligibility re-check | Mandatory on day 1 |
| Form 13- Daily assessments | From day 1 to day 30 |
| Form 14- Change to trial treatment administration | From day 1 to day 30, if indicated on form 13 |
| Form 15- Discontinuation of trial treatment | Mandatory for all consented participants |
| Form 16- Completion of 30 day study observation period | Mandatory for all consented participants |
| Form 17a- Day 60 (+/- 3 days): follow- up assessments | Mandatory for all consented participants who completed the first 30 days (indicated on form 16) |
| Form 17b- Day 120 (+/- 14 days): follow-up assessments | Mandatory for all consented participants who completed the first 60 days (indicated on form 17a) |
| Form 18- Adverse event | From day 1 up to day 60, if applicable |
| Form 19- Safety outcome: thrombotic events or veno occlusive disease | From consent up to study day 120, if applicable |
| Form 20- Health questionnaire: EQ-5D-5L | At randomisation, study day 12 (+/- 2 days), study day 30 (+/-2 days), study day 120 (+/- 14 days) |
| Form 21- Health questionnaire: FACT-Th18 | At randomisation, study day 12 (+/-2 days), study day 30 (+/- 2 days) |
| Form 22a- Health economics | Study day 30 (+/- 2 days) |
| Form 22b- Health economics | Study day 120 (+/-14 days) or last day of follow-up |

# **Statistical Analysis Plan**

Table 2 Trial Schedule (Assessments)

| Trial Assessment | Consent | Days<br>between<br>consent<br>and<br>random-<br>isation | Day R Day of random- isation platelet count ≤ 50x10 <sup>9</sup> /I | Days<br>between<br>Day R and<br>study day<br>1 | Day 1 1st day of trial treatment | Day 2 | Days 3 -<br>11 | Day 12<br>(± 2) | Days 13<br>- 29 | Day 30<br>(± 2) | Day 60<br>(± 3) | Day 120<br>(± 7) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Demographics and medical history | Х | | | | | | | | | | | |
| Eligibility Assessment | Х | | | | X<br>(Prior to<br>starting<br>drug) | | | | | | | |
| Informed consent | Х | | | | | | | | | | | |
| Transfusion requirements | | | Х | Х | Х | Х | Х | Х | х | x | | |
| Bleeding Assessment | | | Х | Х | X | Х | Х | Х | Х | х | | |
| Trial treatment accountability | | | | | Х | Х | Х | Х | х | x | | |
| Quality of life assessment | | | Х | | | | | Х | | х | | x |
| Health economic evaluation | | | | | | | | | | х | | Х |
| Thrombotic<br>Assessment | | Medical<br>notes | Medical<br>notes | Medical<br>notes | Medical<br>notes | Medical<br>notes | Medical<br>notes | Medical<br>notes | Medical<br>notes | Face to face<br>OR<br>Telephone<br>follow-up | | Face to face<br>OR Tele-<br>phone<br>follow-up |
| Highest recorded temperature each day | | | Х | | Х | Х | х | X | Х | | | |
| SAE Assessment | | | | | Х | Х | Х | Х | Х | х | Х | |

# Statistical Analysis Plan

Table 3 Trial Schedule (Investigations)

| Trial Assessment | Consent | Days<br>between<br>consent<br>and<br>randomis-<br>ation | Day R Day of randomisation; platelet count ≤ 50x10 <sup>9</sup> /I | Days<br>between Day<br>R and study<br>day 1 | Day 1<br>1st day<br>of trial<br>treatment | Day 2 | Days 3 -11 | Day 12<br>(± 2) | Days 13 -29 | Day 30<br>(± 2) |
|---|---|---|---|---|---|---|---|---|---|---|
| Pregnancy Test<br>(if applicable) | х | | | | | | | | | |
| Urine dipstick | Х | | | | | | | | | |
| Haemoglobin | X | | x | | X | X | x | x | X | x |
| Platelet count | X | x | x | x | x | x | x | x | x | x |
| Prothrombin<br>Time (or INR if<br>PT not available) | х | | | | | | | | x | |
| Serum creatinine (U&E) | х | | x | | х | х | Required three times a week | X | Required three times a week | х |
| Liver function<br>tests:bilirubin<br>and albumin | х | | x | | | x | Required if<br>VOD is<br>reported 3<br>times a<br>week | x | Required if VOD is reported 3 times a week | |
| HLA Antibody screen† | х | | | | | | | | | |
| | | IN | VESTIGATIONS ON | ILY TO BE PERF | ORMED AT SEL | ECTED PAR | TICIPATING CE | NTRES | | |
| Assays for fibrinolysis | Х | | х | | | х | | | Required three times a week | |

X: measurement required

† HLA Antibodies to be rechecked if participant becomes refractory to platelet transfusions please see section 6.4.1

# Statistical Analysis Plan

# 3.2 Procedures for recording and reporting outcomes

CRFs will be used to collect data from study entry. Two participant identifiers (trial number allocated at consent and initials) will be used on all CRFs. Data will be recorded by electronic data capture (EDC). Prime responsibility for the complete collection of data for each centre will reside with the local Principal Investigator but may be delegated (for example to a research nurse). Overall responsibility for collating data from all centres will reside with the Trial Manager.

#### 3.3 SAE Review

As part of pharmacovigilance procedures, all blinded SAEs will be reviewed by the Chief Investigators in real-time.

#### 3.4 Other assessments

None.

#### 3.5 Trial Data Management and Verification

Quality control of data entered and data cleaning will be performed by the trial data manager and will be detailed in the Data Management Plan (FRM4727). This will include performing range, data completeness and consistency checks. Once this stage is finished, the trial dataset will be declared frozen and exported from the MACRO database for final data review and validation checks by a statistician, who will raise data queries with the trial manager or data manager. Once the trial statistician, data manager, and trial manager are satisfied that all queries have been resolved, the database will be locked. The locked database will be exported to the Statistical Master File and then imported into SAS and used for final analysis.

#### 4. Detailed Analysis Plan

#### 4.1 Interim analysis

Owing to the need to establish both the efficacy and safety of anti-fibrinolytic therapy, the intention is that TREATT will not stop randomising participants if anti-fibrinolytic therapy appears to show effectiveness in an interim analysis. This is because the trial will need to collect additional information on safety endpoints. This is judged important due to the low power the trial has to detect increased rates of thromboembolic events. Because TXA is currently being used off-label in thrombocytopenic participants, it is similarly judged important that any deleterious effect of anti-fibrinolytic therapy with respect to bleeding in thrombocytopenic participants be documented at a level that would be clinically and statistically credible. The Data Monitoring Committee will have overall oversight and can recommend terminating the trial early for these or any other safety concerns.

An interim analysis will be performed after 300 participants have been in the trial for 30 days. A summary of SAEs, UARs, thrombotic events, veno-occlusive disease and death, by treatment arm, will be provided to the Data Monitoring Committee. This summary will be performed by the independent statistician, and will remain inaccessible to the trial statistician, to ensure the trial statistician remains blinded. The population used for safety analyses will be all participants who receive any amount of trial treatment, using data gathered from first administration of trial treatment until up to 120 days after first administration of trial treatment. The population used

# **Statistical Analysis Plan**

for safety analyses of thrombotic events will be all participants who receive any amount of trial treatment, using data gathered from time of consent until 120 days after first administration of trial treatment.

In addition, a multivariate test for heterogeneity of UK and Australian baseline participant characteristics will be performed by the trial statistician. The population used for this analysis will be a modified intention to treat population including all eligible randomised participants whose platelet count falls to 30x109/L or below. Sex, diagnosis (acute leukaemia or not) and treatment plan (autograft or not) will be analysed as binary outcomes. The normal approximation to the binomial will be applied for each binary variable and sex, diagnosis (acute leukaemia or not), treatment plan (autograft or not) and haemoglobin at randomisation will be compared using Hotelling's T-squared test, as long as the following criteria are fulfilled: (i) the estimated proportions are not close to the [0,1] boundaries; (ii) the number of participants in each binary outcome category is > 5; (iii) for each binary variable, 3 standard deviations above and below the expected proportion is within the range [0,1]. If not all the criteria are fulfilled, an alternative test will be considered: a logistic regression of participant country (UK or not) on sex, diagnosis (acute leukaemia or not), treatment plan (autograft or not) and haemoglobin at randomisation will be performed and the concordance statistic and its 95% confidence interval will be calculated. A confidence interval that does not include 0.5 would indicate evidence of a difference between UK and Australian participants. A summary of the multivariate test will be provided to the Data Monitoring Committee. Only strong evidence of a difference between UK and Australian participants will be considered as evidence of heterogeneity. If evidence of heterogeneity between UK and Australian participants is identified in the interim analysis, subgroup analysis by country of participant will be performed for the primary outcome in the main analysis.

#### 4.2 Analysis principles

Unless otherwise specified, all tests will be two-sided and p-values of less than 0.05 will be considered as evidence of a difference between treatment arms.

Multiple comparisons will be performed and this may increase the probability of observing a statistically significant result by chance. No adjustments will be made to account for multiple testing.

P-values will be reported to four decimal places with p-values less than 0.00005 as <0.0001. SAS or R will be used to conduct analyses.

All analyses will be adjusted for the stratification variable (recruitment site). Recruitment site will be accounted for by including a random effect in each model.

All hazard, odds and rate ratios will be presented as active treatment versus placebo. A ratio which is greater than 1 indicates that the hazard, odds or rate is greater in the active treatment arm. 95% confidence intervals will be presented with all ratios. P-values for regression models will be obtained by comparing -2 x log-likelihood values for models with and without the treatment term.

The key demographics and clinical condition of the participants at consent will be presented for each arm of the trial to describe the cohort. A CONSORT diagram will be presented to show how participants progressed through the trial.

# **Statistical Analysis Plan**

### 4.2.1 Efficacy population

The population used for efficacy analyses will be a modified intention to treat population (mITT) including all randomised participants whose platelet count falls to  $30x10^9$ /L or below. Data are gathered for 30 days from the day the first dose of trial treatment is administered or is planned to be administered for those participants who did not receive treatment. Participants will be analysed in the arm that they were randomised to. Randomised participants whose platelet counts do not fall to  $30x10^9$ /L or below will be excluded from the analysis, as will participants who develop exclusion criteria after randomisation and prior to their count falling to  $30x10^9$ /L or below. These exclusions are deemed appropriate as the early randomisation is for pragmatic reasons only. Characteristics of all randomised participants will be compared to the mITT population to ensure that excluded participants are similar across the arms.

Unless otherwise specified, all analyses will be by this mITT. All subjects who fulfil the mITT requirements will be included in the analyses. Subjects whose platelet count falls to  $30x10^9/L$  or below will be included in the analyses, even if they were randomised in error, did not receive trial treatment, stopped trial treatment "early", or received prophylactic transfusions not in accordance with the protocol.

Rationale: Owing to the emergent nature of treatment of thrombocytopenic participants, participants are randomised in a double blind fashion to the treatment arms when platelet levels drop below  $50x10^9$ /L. This will allow time for the pharmacy to prepare the trial treatment, and for the trial treatment to be available when the platelet count falls to  $30x10^9$ /L or below. This has been instituted for pragmatic reasons and will guard against delays in the availability of the trial treatment.

The main outcome analysis will be based on the mITT population. However, a per-protocol analysis of the primary outcome will also be performed. This per-protocol analysis will exclude all participants who were randomised in error and all participants who did not adhere to a set of minimum protocol-adherence criteria during the first 30 days of the trial. The criteria are:

- The participant commenced trial treatment within 72 hours of the first recorded platelet count ≤ 30 x 10<sup>9</sup>/L, OR if the participant was admitted with a platelet count already below 30 x 10<sup>9</sup>/L within 72 hours after the start of chemotherapy or conditioning for a stem cell transplant.
- The participant received trial treatment and only received the trial treatment prescribed to them and did not receive open label tranexamic acid, other antifibrinolytic agent or procoagulant drug
- The participant only received the correct dose of the trial treatment prescribed to them.
- The participant did not receive trial treatment after the point at which discontinuation of trial treatment should have occurred.

Participants who did not meet all the trial eligibility criteria and/or met at least one of the trial exclusion criteria will be considered as randomised in error. Participants who were randomised in error and received study intervention will be considered a protocol deviation. Participants who withdrew from the trial after starting trial treatment, who missed a dose of trial treatment or who chose to stop trial treatment "early" *are* included in the per protocol analysis.

### 4.2.2 Safety population (apart from thrombotic events)

The population used for safety analyses will be all participants who receive any amount of trial treatment, using data gathered from first administration of trial treatment until up to 120 days after first administration of trial treatment.

#### 4.2.3 Thrombotic Event Safety population

# **Statistical Analysis Plan**

The population used for safety analyses of thrombotic events will be all participants who receive any amount of trial treatment, using data gathered from time of consent until 120 days after first administration of trial treatment.

#### 4.3 Analysis of primary outcome measures

### Primary efficacy analysis

The proportion of participants who die or have bleeding of grade 2 or above by WHO criteria during the first 30 days from the day the first dose of trial treatment is administered, will be estimated by the Kaplan-Meier method and compared by treatment arm using Cox regression analysis. All participants whose platelet count dropped to  $30x10^9$ /L or below, regardless of length of follow-up will be included. Participants withdrawn or lost to follow up before day 30 will be censored at the time that they withdrew/were lost to follow up. Any missing bleeding assessments during the 30-day follow up period or to the last point of contact, whichever is first, will be assumed to be grade 1 or below.

If there is evidence of a difference in the primary outcome between treatment arms, the number needed to treat (NNT) (for benefit) will be presented. NNT is the number of participants who need to be treated with tranexamic acid in addition to standard care in order for one additional participant to benefit. It is calculated as 1 / (difference in proportion experiencing the primary outcome in each treatment arm as a decimal).

### 4.4 Analysis of secondary outcome measures

#### Secondary efficacy outcomes

- Proportion of days with bleeding up to study day 30 will be compared by treatment arm
  using binary logistic regression analysis (bleeding or not on any given day). Correlation
  at participant level will be accounted for by including a random participant effect.
- Time to first episode of bleeding of WHO grade 2 or greater up to study day 30 will be estimated using the cumulative incidence function, with the competing risk of death prior to bleeding of WHO grade 2 or greater. Median, IQR will be reported by treatment arm. To accommodate a random centre effect, Cox regression analysis will be used to compare time to first episode of bleeding of WHO grade 2 or greater between treatment arms. Participants who have not experienced bleeding of WHO grade 2 or greater will be censored at day 30 or at the point of last contact, whichever is first. Participants who died prior to study day 30 and did not experience bleeding of WHO grade 2 or greater will be censored at the time of death. The estimate of the hazard of bleeding of WHO grade 2 or greater from this model should be interpreted with caution because it does not properly account for the competing risk of death. However, since the number of deaths are predicted to be small, the impact of the competing risk is likely to be negligible. This will be explored by examining the cumulative incidence function for death prior to bleeding of WHO grade 2 or greater.
- Highest grade of bleeding up to study day 30 will be compared by treatment arm using an ordinal logistic regression model, modelling grade as an ordinal categorical outcome.
- Number of platelet transfusions/participant up to study day 30 will be compared by treatment arm using a negative binomial model. The model will include an offset to account for the number of days the participant spent in hospital, up to 30 days or to the last point of contact, whichever is first. In addition, unadjusted median, IQR number of platelet transfusions per day in hospital will be reported.
- Number of red cell transfusions/participant up to study day 30 will be compared by treatment arm using a negative binomial model. The model will include an offset to account for the number of days the participant spent in hospital, up to 30 days. In addition,

# **Statistical Analysis Plan**

- unadjusted median, IQR number of red cell transfusions per day in hospital will be reported.
- Proportion of participants surviving up to 30 days without a platelet transfusion will be estimated by the Kaplan-Meier method and compared by treatment arm using Cox regression analysis. The event of interest is time to first platelet transfusion or death. Participants withdrawn or lost to follow up before day 30 will be censored at the time that they withdrew/were lost to follow up.
- Proportion of participants surviving up to 30 days without a red cell transfusion will be estimated by the Kaplan-Meier method and compared by treatment arm using Cox regression analysis. The event of interest is time to first red cell transfusion or death. Participants withdrawn or lost to follow up before day 30 will be censored at the time that they withdrew/were lost to follow up.
- Quality of life at study days 12 and 30 will be assessed using FACT-G and FACT-Th health questionnaires. For the FACT-G subscale scores (physical well-being, social/family well-being, emotional well-being, functional well-being), FACT-G total score and FACT-Th total score, mean (SD) will be calculated and compared by treatment arm using normal regression analysis. For each normal linear regression model, residual plots will be examined. If there is substantial evidence of skew or non-constant variance, log-transformed values will be used instead.

#### Safety outcomes

- Number of thrombotic events from first administration of trial treatment up to and including 120 days after the first dose of trial treatment is received, per day at risk, will be described by arm.
- Number of participants developing Veno-occlusive Disease (VOD; Sinusoidal obstructive syndrome, SOS) within 60 days of first administration of trial treatment, will be described by arm.
- All-cause mortality during the first 30 days and 120 days after the first dose of trial treatment is administered will be estimated by the Kaplan-Meier method and compared using Cox regression analysis. Participants withdrawn or lost to follow up before day 30/day 120 will be censored at the time that they withdrew/were lost to follow up.
- Death due to thrombosis during the first 120 days after the first dose of trial treatment is administered will be estimated using the cumulative incidence function, with the competing risk of death due to other causes. To accommodate a random centre effect, Cox regression analysis will be used to compare death due to thrombosis between treatment arms. Participants who have not died will be censored at day 120 or at the point of last contact, whichever is first. Participants who died prior to day 120 from other causes will be censored at the time of death. If numbers of deaths due to thrombosis are very small, the number of deaths will simply be described by arm.
- Death due to bleeding during the first 30 days after the first administration of trial treatment is received will be estimated using the cumulative incidence function, with the competing risk of death due to other causes. To accommodate a random centre effect, Cox regression analysis will be used to compare death due to bleeding between treatment arms. Participants who have not died will be censored at day 120 or at the point of last contact, whichever is first. Participants who died prior to day 120 from other causes will be censored at the time of death. If numbers of deaths due to bleeding are very small, the number of deaths will simply be described by arm.
- Number of serious adverse events from first administration of trial treatment until 60 days
  after the first dose of trial treatment is administered, per day at risk, will be summarised
  by arm, including number of symptomatic thrombotic events (venous thromboembolisms
  and arterial ischaemic events), veno-occlusive disease, sepsis, organ failure and deaths.

# **Statistical Analysis Plan**

#### 4.5 Other outcome measures

 Proportion of days with thrombocytopenia (platelet count <10x10<sup>9</sup>/L) from consent up to study day 30 will be compared by treatment arm using binary logistic regression analysis (thrombocytopenic or not on any given day). Correlation at participant level will be accounted for by including a random participant effect. If the number of thrombotic events is very small, the proportions will simply be described by arm.

- Proportion of days with thrombocytopenia (platelet count <30x10<sup>9</sup>/L) from consent up to study day 30 will be compared by treatment arm using binary logistic regression analysis (thrombocytopenic or not on any given day). Correlation at participant level will be accounted for by including a random participant effect. If the number of thrombotic events is very small, the proportions will simply be described by arm.
- Proportion of days with thrombocytopenia (platelet count <50x10<sup>9</sup>/L) from consent up to study day 30 will be compared by treatment arm using binary logistic regression analysis (thrombocytopenic or not on any given day). Correlation at participant level will be accounted for by including a random participant effect. If the number of thrombotic events is very small, the proportions will simply be described by arm.
- Proportion of days with fever (highest daily temperature ≥ 38.1°C) of days spent in hospital, up to study day 30, will be analysed using binary logistic regression analysis (fever or not on any given day). Correlation at participant level will be accounted for by including a random participant effect.
- Reasons for platelet and red cell transfusions will be described by arm.
- A plot depicting median, IQR platelet count over time from consent up to study day 30, by arm, will be produced. Where consent, randomisation and/or treatment occurred on the same day, the participant's platelet count will only be included in the median calculation for the last of the concurrent events.
- A plot depicting overall survival from randomisation up to study day 120, by arm, will be produced.
- Trial treatment will be summarised by arm, including number of participants who
  changed route or frequency, number of participants who missed a dose, reasons for
  discontinuation of treatment. Median, IQR number of days on trial treatment and on oral
  trial treatment, from the first day of treatment administration until discontinuation of trial
  treatment, for participants who received at least one dose of trial treatment, will be
  estimated using competing risks analysis. Death prior to discontinuation of trial
  treatment will be considered as the competing risk.
- Number of granulocyte transfusions/participant up to study day 30 will be summarised by treatment arm.
- Location of bleeding up to study day 30 will be summarised, by treatment arm
- Number of participants requiring interventions and procedures for bleeding up to study day 30 will be summarised by treatment arm. This may be sub-categorised by type of intervention or procedure if there are large numbers of participants requiring interventions and procedures.
- Number of participants requiring concomitant medication (categorised as medication increasing risk of bleeding, medication decreasing risk of bleeding, no concomitant medication) up to study day 30 will be summarised by treatment arm. This may be subcategorised by type of concomitant medication if there are large numbers of participants requiring concomitant medication.
- Number of participants on Mylotarg during the first 30 days of the trial will be summarised by treatment arm.

# Statistical Analysis Plan

# 4.6 Sub-Group analyses

Subgroup analyses will be performed for the primary outcome in the main analysis by including an interaction term. Analysis will be performed using the same methods as for the primary outcome, except a covariate and treatment-covariate interaction will be included in the model for each of the following variables in turn:

- Country of participant (UK vs. Australia), if evidence of heterogeneity between UK and Australian participants is identified in the interim analysis
- Platelet count at consent (≤30x10<sup>9</sup>/L vs. >30x10<sup>9</sup>/L)

Treatment compliance during first 30 days of the trial (participant decided to stop taking trial treatment vs. participant did not decide to stop taking trial treatment). Although participants may decide to stop taking trial treatment for many reasons, the main reason is thought to be an unwillingness to take the large, over-encapsulated oral trial treatment. The over-encapsulated oral trial treatment is to be replaced with smaller tablets in the UK and Australia. Therefore, an additional analysis of treatment compliance will be performed using four mutually-exclusive categories: participant decided to stop taking trial treatment during the period of over-encapsulated oral treatment; participant decided to stop taking trial treatment during the period of over-encapsulated oral treatment as tablets; participant did not decide to stop taking trial treatment during the period of over-encapsulated oral treatment; participant did not decide to stop taking trial treatment during the period of oral treatment as tablets. The number of UK participants who discontinued IV trial treatment during the period in September 2018 when oral treatment was unavailable will be described by arm.

### 4.7 Sensitivity analyses

- The key demographics and clinical condition of participants at consent will be described for each arm of the trial, comparing all randomised participants with the mITT population to ensure that excluded participants are similar across the arms.
- Per-protocol analysis of the primary outcome. This analysis will exclude all participants who did not adhere to a set of minimum protocol-adherence criteria during the first 30 days of the trial. Participants who were randomised in error will be excluded from this analysis. The per-protocol analysis will be performed using the same method as for the mITT analysis. Protocol-adherence will be summarised by treatment arm. In addition, since the per-protocol analysis may lead to an over-estimation of the difference in the proportion experiencing the primary outcome in each treatment arm, which may be explained by differing levels of protocol-adherence in each treatment arm, an instrumental variable analysis will be performed. The randomisation arm will be used as the instrument. The instrumental variable estimate will be calculated as the mITT estimate of the difference in the proportion experiencing the primary outcome in each treatment arm / proportion adhering to the minimum compliance criteria in the active treatment arm. The standard error of the instrumental variable estimate will be calculated using two-stage least squares.
- Some participants may withdraw or be lost to follow up during the conduct of the trial. In addition, some participants who are followed up for the full 30 days may be missing some bleeding assessments. In these cases, it is impossible to know whether such participants would be either less or more likely to experience bleeding if they had complete bleeding assessments for the full 30-day follow up period. Sensitivity of the primary outcome to incomplete follow up and missing bleeding assessments will be assessed by re-calculating the primary outcome, by arm, for all participants included in the mITT analysis, after imputing all missing bleeding assessments up to study day 30.

# Statistical Analysis Plan

Imputation will be performed using multiple imputation by fully conditional specification (Van Buuren, 2007), with the number of imputations equal to the percentage of missing data.

- Number of days between platelet count first 30 x 10<sup>9</sup>/L or below OR if the participant was admitted with a platelet count already below 30 x 10<sup>9</sup>/L, number of days between the start of chemotherapy or conditioning for a stem cell transplant, and start of trial treatment, or planned start for those participants who did not receive treatment, will be summarised by treatment arm, for all participants included in the mITT analysis. It is important to monitor this since the 30-day analysis period only begins at the start of study treatment.
- Number of bleeds between platelet count first 30 x 10<sup>9</sup>/L or below and start of trial treatment or planned start for those participants who did not receive treatment will be summarised by treatment arm, for all participants included in the mITT analysis. It is important to monitor whether any bleeds occurred prior to the start of the 30-day analysis period.

### 4.8 Procedures for handling Missing Data

For all outcomes, the volume of missing data will be summarised by treatment arm.

Participants withdrawn or lost to follow up before day 30 will be included in the primary outcome analysis (and in secondary outcome analyses where possible), censoring at the time that they withdrew/were lost to follow up.

It is expected that deaths and other safety outcomes, other than for participants withdrawn or lost to follow up, will be fully reported.

For the main analysis of the primary outcome, any missing bleeding assessments during the 30-day follow up period or to the last point of contact, whichever is first, will be assumed to be grade 1 or below. Sensitivity of the primary outcome to missing data will be assessed as per the sensitivity analysis described above.

Missing values for secondary and baseline characteristics will not be imputed. Missing data will be excluded from the relevant analyses.

#### 5. Data Analysis Tables to be Completed

Data analysis will be based on the following tables.

#### 5.1 Interim analysis tables

Table 1 Baseline characteristics for UK vs. Australian participants – data are number (%) for categorical variables, and mean (SD) for continuous variables

| | UK (n=) | Australia<br>(n=) | P value |
|----------------------------|---------|-------------------|---------|
| Sex: Male | | | |
| Diagnosis: Acute leukaemia | | | |
| Treatment plan: Autograft | | | |
| Haemoglobin at | | | |
| randomisation (G/L) | | | |

<sup>&#</sup>x27;Other' diagnosis includes xxx and 'other' treatment plan includes xxx.

Sex is missing for xxx participants, of which xxx are not available.

Diagnosis is missing for xxx participants, of which xxx are not available.

Treatment plan is missing for xxx participants, of which xxx are not available.

Haemoglobin at randomisation is missing for xxx participants, of which xxx are not available.

# **Statistical Analysis Plan**

Table 2 Safety data summary - data are numbers

| Outcome | Arm A<br>(n=) | Arm B<br>(n=) | Overall (n=) |
|---|---|---|---|
| Total number of serious adverse events (SAE) up to day 60 | | | |
| Sepsis | | | |
| Organ failure | | | |
| GvHD | | | |
| Transfusion reaction | | | |
| Fever | | | |
| Other SAEs | | | |
| Number of participants experiencing at least one SAE | | | |
| Symptomatic thrombotic events up to day 120 | | | |
| Venous thromboembolisms | | | |
| Arterial ischaemic events | | | |
| Veno-occlusive disease up to day 120 | | | |
| Unexpected adverse reactions up to day 60 | | | |
| Deaths up to day 120 | | | |

# **Statistical Analysis Plan**

# 5.2 Screening, Recruitment and Follow-up tables

# 5.2.1 Recruitment by Centre

# Table xx Recruitment by centre

| Centre | Number of participants screened | Number of eligible participants | %<br>eligible<br>of those<br>screened | Number of participants approached | Number of participants consented | Number of randomisations | %<br>randomised<br>of those<br>eligible |
|---|---|---|---|---|---|---|---|
| Birmingham Heartlands Hospital | | | | | | | |
| Derriford Hospital, Plymouth | | | | | | | |
| Kings College Hospital, London | | | | | | | |
| Churchill Hospital, Oxford | | | | | | | |
| Freeman Hospital, Newcastle | | | | | | | |
| University Hospital, Coventry | | | | | | | |
| St James's Hospital, Leeds | | | | | | | |
| Bristol Haematology & Oncology<br>Centre | | | | | | | |
| Victorian Comprehensive Cancer<br>Centre (formerly Peter<br>MacCallum Cancer Centre),<br>Melbourne, | | | | | | | |
| St. Vincent's Hospital, Melbourne | | | | | | | |
| The Beatson Oncology Centre,<br>Glasgow | | | | | | | |
| Royal Adelaide Hospital | | | | | | | |

# **Statistical Analysis Plan**

| | 1 | _ | 1 |
|------------------------------------------------------|---|---|---|
| The Alfred Hospital, Melbourne | | | |
| Andrew Love Cancer Centre,<br>Barwon Health, Geelong | | | |
| Salisbury District Hospital, UK | | | |
| Royal Devon and Exeter Hospital | | | |
| University College London<br>Hospital | | | |
| Lincoln County Hospital | | | |
| Belfast City Hospital | | | |
| Queen Elizabeth Hospital,<br>Birmingham | | | |
| Royal United hospital, Bath | | | |
| Royal North Shore Hospital,<br>Sydney | | | |
| Westmead Hospital, Sydney | | | |
| Canberra Hospital | | | |
| St Vincent's, Sydney | | | |

# **Statistical Analysis Plan**

# Table xx Participants withdrawn

| Participant ID | Arm | Reason for withdrawal | Stage of withdrawal |
|----------------|-----|-----------------------|---------------------|

### 5.2.3 Participants randomised in error

# Table xx Participants randomised in error

| Participant ID | Arm | Detail of error |
|----------------|-----|-----------------|

5.2.4 Participants entered in trial more than once (if relevant) or co-enrolled in other trials

### Table xx Participants co-enrolled in other trials

| Participant ID | Arm | Detail of co-enrolment |
|----------------|-----|------------------------|

### 5.2.5 Protocol Deviations

### Table xx Protocol deviations

| Participant ID | Arm | Detail of protocol deviation |
|----------------|-----|------------------------------|

# 5.3 Baseline Characteristics tables

# Table xx Baseline characteristics- data are number (%) for categorical variables, and mean (SD) for continuous variables

| Active arm | Placebo arm | Overall (n=) |
|------------|-------------|--------------|
| (n=) | (n=) | |

# Statistical Analysis Plan

| Male | |
|---------------------------------|------|
| Age (years) | |
| Ethnicity | |
| White | |
| Asian | |
| Black African | |
| Black Caribbean | |
| Arab/other Middle East ancestry | |
| Aboriginal | |
| Other | |
| Mixed ethnic group: | |
| White/Black Caribbean | |
| White/Black African | |
| White/Asian | |
| White/Aboriginal | |
| White/Other | |
| Other mixed ethnic group | |
| Height (cm) | |
| Weight (kg) | |
| Diagnosis | |
| AML | |
| ALL | |
| APL | |
| CML | |
| CLL | |
| Hodgkins Lymphoma | |
| Non-Hodgkins Lymphoma | |
| Myeloma | |
| MDS | |
| Other | |
| Treatment plan | <br> |
| Induction chemotherapy | |
| Consolidation chemotherapy | |
| Autograft | |
| Allograft | |
| Other | |
| Platelet count at consent | |
| (x 10 <sup>9</sup> /L) | |
| Platelet count at randomisation | |
| (x 10 <sup>9</sup> /L) | |
| Haemoglobin at consent (G/L) | |
| Haemoglobin at randomisation | |
| (G/L) | |
| FACT-G subscale score at | |
| randomisation | |
| Physical well-being | |
| Social/family well-being | |
| Emotional well-being | |
| Functional well-being | |
| FACT-G total score at | |
| randomisation | |

# Statistical Analysis Plan

| FACT-Th total score at randomisation |
|--------------------------------------|
| Medical history |
| Diabetes requiring treatment |
| Hypertension requiring |
| treatment |
| Renal impairment requiring |
| treatment |
| Confirmed invasive fungal |
| infection |
| Other malignancy |
| HLA antibodies |

<sup>&#</sup>x27;Other' diagnoses were xxx and 'other' treatment plans were xxx.

#### 5.4 Primary Outcome table(s)

#### Table xx Primary outcome table

| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) | P value |
|---|---|---|---|---|
| Proportion of participants<br>who die or have bleeding of<br>WHO grade 2 or above from<br>day 1 up to study day 30 - %<br>(95% CI) | | | | |
| Hazard ratio (95% CI) | | | | |
| Risk difference (95% CI) | | | | |
| Number needed to treat <sup>1</sup> – N | | | | |
| Proportion of missing bleeding assessments from day 1 up to study day 30 – n/N (%) | | | | |
| Proportion of participants<br>missing vital status at study day<br>30 – n/N (%) | | | | |
| All primary outcome analyses are ad | • | ntre. | | |

#### Secondary Outcome table(s) 5.5

#### Table xx Secondary efficacy outcomes table

| Outcome | Active arm (n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) | P value |
|---|---|---|---|---|
| Proportion of days with WHO grade 2 bleeding or above – % (95% CI) | | (***/ | | |
| Odds ratio <sup>1</sup> (95% CI) | | | | |

# Statistical Analysis Plan

| Time to first episode of bleeding | |
|-------------------------------------------|---|
| of WHO grade 2 or greater (days) | |
| (median <sup>2</sup> , IQR <sup>2</sup> ) | |
| Hazard ratio (95% CI) | |
| Highest grade of bleeding a | |
| participant experiences | |
| Grade 0 – n/N (%) | |
| Grade 1 – n/N (%) | |
| Grade 2 – n/N (%) | |
| Grade 3 – n/N (%) | |
| Grade 4 – n/N (%) | |
| Grade unassigned – n/N (%) | |
| Proportional odds ratio (95% CI) | |
| Grades 2, 3 or 4 – n/N (%) | |
| Number of platelet | |
| transfusions/participant (units) | |
| up to study day 30 (median, IQR) | |
| Rate ratio (95% CI) | |
| Number of red cell | |
| transfusions/participant (units) | |
| up to study day 30 (median, IQR) | |
| Rate ratio (95% CI) | , |
| Proportion of participants | |
| surviving up to 30 days without | |
| a platelet transfusion – % (95% | |
| CI) | |
| Hazard ratio (95% CI) | |
| Proportion of participants | |
| surviving up to 30 days without | |
| a red cell transfusion – % (95% | |
| CI) | |
| Hazard ratio (95% CI) | |

#### Table xx **Quality of life**

| Outcome | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) | P-value |
|---|---|---|---|---|
| FACT-G subscale score at study day 12 | | | | |
| Physical well-being - mean (SD) | | | | |
| Social/family well-being - mean (SD) | | | | |
| Emotional well-being - mean (SD) | | | | |
| Functional well-being - mean (SD) | | | | |

All secondary efficacy outcome analyses are adjusted for centre.

<sup>1</sup> Odds ratio from logistic regression model, also adjusted for participant.

<sup>2</sup> Lower quartile will be reported. Median and upper quartile will be reported if achieved.

# **Statistical Analysis Plan**

| FACT-G total score at study day 12 - mean (SD) | | | | |
|---|---|---|---|---|
| FACT-Th total score at study day 12 - mean (SD) | | | | |
| FACT-G subscale score at study day 30 | | | | |
| Physical well-being - mean (SD) | | | | |
| Social/family well-being - mean (SD) | | | | |
| Emotional well-being - mean (SD) | | | | |
| Functional well-being - mean (SD) | | | | |
| FACT-G total score at study day 30 - mean (SD) | | | | |
| FACT-Th total score at study day 30 - mean (SD) | | | | |
| All quality of life outcome analyses are adjusted for | or centre. | • | • | • |

# Table xx Safety outcomes table

| | Active arm | Placebo<br>arm | Overall<br>(n=) | P value |
|---|---|---|---|---|
| Outcome | (n=) | (n=) | | |
| All-cause mortality during the first 30 | | | | |
| days after the first dose of trial treatment | | | | |
| is administered – % (95% CI) | | | | |
| Hazard ratio (95% CI) | | | | |
| All-cause mortality during the first 120 | | | | |
| days after the first dose of trial treatment | | | | |
| is administered – % (95% CI) | | | | |
| Hazard ratio (95% CI) | | | | |
| Number of thrombotic events from first | | | | |
| administration of trial treatment up to and | | | | |
| including 120 days after the first dose of | | | | |
| trial treatment is received, per day at risk | | | | |
| (N) | | | | |
| Number of participants developing Veno- | | | | |
| occlusive Disease within 60 days of first | | | | |
| administration of trial treatment (N) | | | | |
| Death due to thrombosis during the first | | | | |
| 120 days after the first dose of trial | | | | |
| treatment is administered – % (95% CI) | | | | |
| Hazard ratio (95% CI) | | 1 | | |
| Death due to bleeding during the first 30 | | | | |
| days after the first administration of trial | | | | |
| treatment is received – % (95% CI) | | | | |
| Hazard ratio (95% CI) | | | | |

# Table xx Safety data summary - data are numbers

# Statistical Analysis Plan

| Outcome | Active arm (n=) | Placebo<br>arm (n=) | Overall<br>(n=) |
|---|---|---|---|
| Total number of serious adverse events (SAE) up to day 60 | | | |
| Sepsis | | | |
| Organ failure | | | |
| GvHD | | | |
| Transfusion reaction | | | |
| Fever | | | |
| Other SAEs | | | |
| Number of participants experiencing at least one SAE | | | |
| Symptomatic thrombotic events up to day 120 | | | |
| Venous thromboembolisms | | | |
| Arterial ischaemic events | | | |
| Veno-occlusive disease up to day 120 | | | |
| Unexpected adverse reactions up to day 60 | | | |
| Deaths up to day 120 | | | |

All SAEs, unexpected adverse reactions, thrombotic events and veno-occlusive disease are reported in full in Appendix 1.

# 5.6 Missing Data tables

# Table xx Missing secondary efficacy outcomes data table – n/N (%)

| | Active arm (n=) | Placebo<br>arm (n=) | Overall (n=) |
|---|---|---|---|
| Missing data for platelet transfusions up to study day 30 | | | |
| Missing data for red cell transfusions up to study day 30 | | | |
| Missing data for FACT-G subscale score at study day 12 | | | |
| Missing data for FACT-G total score at study day 12 | | | |
| Missing data for FACT-Th total score at study day 12 | | | |
| Missing data for FACT-G subscale score at study day 30 | | | |
| Missing data for FACT-G total score at study day 30 | | | |
| Missing data for FACT-Th total score at study day 30 | | | |

# **Statistical Analysis Plan**

# 5.7 Other Outcome summary tables

# Table xx Proportion of days with thrombocytopenia

| Outcome | Active arm (n=) | Placebo arm (n=) | Overall (n=) | P value |
|---|---|---|---|---|
| Proportion of days with thrombocytopenia (<10x10 <sup>9</sup> /L) from randomisation up to study day 30 - % (95% CI) | | | | |
| Odds ratio (95% CI) | | | | |
| Proportion of days with thrombocytopenia (<30x10 <sup>9</sup> /L) from randomisation up to study day 30 - % (95% CI) | | | | |
| Odds ratio (95% CI) | | | | |
| Proportion of days with thrombocytopenia (<50x10 <sup>9</sup> /L) from randomisation up to study day 30 - % (95% CI) | | | | |
| Odds ratio (95% CI) | | | | |
| Proportion of missing platelet counts from randomisation up to study day 30 – n/N (%) | | | | |
| All analyses are adjusted for centre and par | ticipant. | | | |

# Table xx Proportion of days with fever

| Outcome | Active arm (n=) | Placebo arm (n=) | Overall (n=) | P value |
|---|---|---|---|---|
| Proportion of days with fever (highest daily temperature ≥ 38.1°C) of days spent in hospital, up to study day 30 - % (95% CI) | | | | |
| Odds ratio (95% CI) | | | | |
| Missing fever data up to study day 30 – n/N (%) | | | | |
| All analyses are adjusted for centre and pa | rticipant. | | | • |

# Table xx Reasons for transfusions – n/N (%)

| Outcome | Active arm (n=) | Placebo<br>arm<br>(n=) | Overall (n=) |
|---|---|---|---|
| Reasons for platelet transfusions | | | |
| Prophylaxis for platelet count ≤10x10 <sup>9</sup> /L | | | |
| Prophylaxis and platelet count >10x10 <sup>9</sup> /L | | | |
| Invasive procedure | | | |
| Active bleeding | | | |

# **Statistical Analysis Plan**

| Missing data for reasons for platelet transfusions |
|----------------------------------------------------|
| Reasons for red cell transfusions |
| Low haemoglobin |
| Active bleeding |
| Other |
| Missing data for reasons for red cell |
| transfusions |

# Table xx Summary of trial treatment

| | Arm A (n=) | Arm B (n=) | Overall (n=) |
|---|---|---|---|
| Number of participants ever on treatment – n/N (%) | | | \ |
| Number of days on treatment – median (IQR) | | | |
| Number of participants ever on oral treatment – n/N (%) | | | |
| Number of days on oral treatment – median (IQR) | | | |
| Number of participants who changed route or frequency (N only)* From oral to IV From IV to oral Reduced frequency Increased frequency Reason for frequency change <sup>1</sup> Renal impairment Other Missing data for route or frequency change – n/N (%) | | | |
| Number of participants who have missed a dose in a 24 hour period – n/N (%) | | | |
| Number of participants who have discontinued treatment – n/N (%) >30 days since started treatment Spontaneous increase in platelet count >50 x 109/L 3 consecutive days with morning platelet count >30 x109/L Received open label TXA, other antifibrinolytic agent or procoagulant drug Started anticoagulant or antiplatelet therapy Visible haematuria Diagnosis of thrombosis Anuric | | | |

# **Statistical Analysis Plan**

| Developed sinusoidal obstructive syndrome Clinical decision Unacceptable adverse reaction to trial treatment |
|---|
| Change in participant's condition |
| Participant's decision |
| Missing data for reason for |
| discontinuation of treatment – n/N (%) |

# Table xx Location of bleeding - n/N (%)

| Location of bleeding | Active arm (n=) | Placebo<br>arm<br>(n=) | Overall (n=) |
|---|---|---|---|
| Skin | | | |
| Oropharyngeal | | | |
| Epistaxis | | | |
| Gastrointestinal | | | |
| Blood in urine | | | |
| Soft tissue and musculoskeletal | | | |
| Haemoptysis | | | |
| Invasive procedure | | | |
| Abnormal vaginal bleeding | | | |
| Retinal or vitreous | | | |
| Body cavity/other | | | |
| Subconjunctiva of the eye | | | |

# Table xx Other outcomes – n/N (%)

| Outcome | Active arm (n=) | Placebo<br>arm<br>(n=) | Overall (n=) |
|---|---|---|---|
| Number of participants on | | | |
| Mylotarg up to study day 30 | | | |
| Missing Mylotarg data up to study | | | |
| day 30 | | | |
| Number of granulocyte | | | |
| transfusions/participant up to | | | |
| study day 30 | | | |
| Missing granulocyte transfusion data | | | |
| up to study day 30 | | | |
| Number of participants requiring | | | |
| interventions and procedures for | | | |
| bleeding up to study day 30 | | | |
| Missing data for interventions and | | | |
| procedures for bleeding up to study | | | |
| day 30 | | | |

<sup>\*</sup> Participants may appear more than once

<sup>&</sup>lt;sup>1</sup> Reason for frequency change not reported for 1 participant.

# **Statistical Analysis Plan**

| Number of participants requiring concomitant medication up to study day 30 |
|---|
| Missing data for concomitant medication up to study day 30 |

# 5.8 Sub-group analysis tables

**Table xx Primary outcome - UK participants vs Australian participants** [table will only be produced if evidence of heterogeneity at the interim analysis]

| | UK | | Australia | |
|---|---|---|---|---|
| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) |
| Proportion of participants who die or have bleeding of WHO grade 2 or above from day 1 up to study day 30 - n/N (%) | | | | |
| Hazard ratio (95% CI) | | | | |
| P-value for interaction term | | | | |
| All primary outcome analyses are adj | justed for ce | ntre. | | |

# Table xx Primary outcome - Platelet count at consent (≤30x109/L vs. >30x109/L)

| | ≤30x10 <sup>9</sup> /L | | >30x | 10 <sup>9</sup> /L |
|---|---|---|---|---|
| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) |
| Proportion of participants<br>who die or have bleeding of<br>WHO grade 2 or above from<br>day 1 up to study day 30 - n/N<br>(%) | | | | |
| Hazard ratio (95% CI) | | | | |
| P-value for interaction term | | | | |
| All primary outcome analyses are ad | justed for cer | ntre. | | |

Table xx\_a Primary outcome - Treatment compliance during first 30 days of the trial (participant decided to stop taking trial treatment vs. participant did not decide to stop taking trial treatment)

| Participant decided to | Participant did not |
|------------------------|----------------------|
| stop trial treatment | decide to stop trial |
| | treatment |

# **Statistical Analysis Plan**

| | Active arm (n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) |
|---|---|---|---|---|
| Proportion of participants who die or have bleeding of WHO grade 2 or above from day 1 up to study day 30 - n/N (%) | | | | |
| Hazard ratio (95% CI) | | | | |
| P-value for interaction term | | | | |
| All primary outcome analyses are adjusted for centre. | | | | |

Table xx\_b Primary outcome - Treatment compliance during first 30 days of the trial (participant decided to stop taking trial treatment during the period of over-encapsulated oral treatment; participant decided to stop taking trial treatment during the period of oral treatment as tablets; participant did not decide to stop taking trial treatment during the period of over-encapsulated oral treatment; participant did not decide to stop taking trial treatment during the period of oral treatment as tablets)

| | decide<br>trial tr<br>duri<br>period<br>encap | cipant<br>d to stop<br>eatment<br>ng the<br>of over-<br>sulated<br>eatment | decide<br>takir<br>trea<br>duri<br>period<br>treatr | icipant d to stop ng trial tment ng the d of oral ment as blets | not de<br>stop ta<br>trea<br>duri<br>period<br>encap | ipant did<br>ecide to<br>king trial<br>tment<br>ng the<br>of over-<br>osulated<br>eatment | not do<br>stop ta<br>trea<br>duri<br>perioo<br>treatr | pant did<br>ecide to<br>king trial<br>tment<br>ng the<br>d of oral<br>ment as<br>olets |
|---|---|---|---|---|---|---|---|---|
| | Active arm (n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) |
| Proportion of participants who die or have bleeding of WHO grade 2 or above from day 1 up to study day 30 - n/N (%) | | | | | | | | |
| Hazard ratio (95% CI) | | | | | | | | |
| P-value for interaction term | | | | | | | | |
| All primary outcome a | nalyses ar | e adjusted | for centre | ). | | | | |

# **Statistical Analysis Plan**

### 5.9 Sensitivity and missing data analysis tables

Table xx Baseline characteristics for all randomised participants vs. all randomised participants with platelet count ≤30x10<sup>9</sup>/L – data are number (%) for categorical variables, and mean (SD) for continuous variables

| | Randomised participants | | Randoı<br>partici<br>with plate<br>≤30x1 | pants<br>let count<br> 0 <sup>9</sup> /L |
|---|---|---|---|---|
| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Active arm (n=) | Placebo<br>arm<br>(n=) |
| Male | | | | |
| Age (years) | | | | |
| Ethnicity | | | | |
| White | | | | |
| Asian | | | | |
| Black African | | | | |
| Black Caribbean | | | | |
| Arab/other Middle East | | | | |
| ancestry | | | | |
| Aboriginal | | | | |
| Other | | | | |
| Mixed ethnic group: | | | | |
| White/Black Caribbean | | | | |
| White/Black African | | | | |
| White/Asian | | | | |
| White/Aboriginal | | | | |
| White/Other | | | | |
| Other mixed ethnic group | | | | |
| Height (cm) | | | | |
| Weight (kg) | | | | |
| Diagnosis | | | | |
| AML | | | | |
| ALL | | | | |
| APL | | | | |
| CML | | | | |
| CLL<br>Haddking Lymphome | | | | |
| Hodgkins Lymphoma | | | | |
| Non-Hodgkins Lymphoma | | | | |
| Myeloma | | | | |
| MDS | | | | |
| Other Treatment plan | | | + | |
| Treatment plan | | | | |
| Induction chemotherapy | | | | |
| Consolidation chemotherapy | | | | |
| Autograft | | | | |
| Allograft | | | | |
| Other | | | | |
| Platelet count at consent | | | | |
| (x 10 <sup>9</sup> /L) | | | | |

# **Statistical Analysis Plan**

| Platelet count at randomisation |
|---------------------------------|
| (x 10 <sup>9</sup> /L) |
| Haemoglobin at consent (G/L) |
| Haemoglobin at randomisation |
| (G/L) |
| FACT-G subscale score at |
| randomisation |
| Physical well-being |
| Social/family well-being |
| Emotional well-being |
| Functional well-being |
| FACT-G total score at |
| randomisation |
| FACT-Th total score at |
| randomisation |
| Medical history |
| Diabetes requiring |
| treatment |
| Hypertension requiring |
| treatment |
| Renal impairment requiring |
| treatment |
| Confirmed invasive fungal |
| infection |
| Other malignancy |
| HLA antibodies |

# Table xx Per protocol analysis

| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) | P value |
|---|---|---|---|---|
| Proportion of participants<br>who die or have bleeding of<br>WHO grade 2 or above from<br>day 1 up to study day 30 - n/N<br>(%) | | | | |
| Hazard ratio (95% CI) | | | | |
| Risk difference (95% CI) | | | | |
| Protocol adherence <sup>1</sup> – n/N (%) | | | | |
| Risk difference <sup>2</sup> (95% CI) – instrumental variable analysis | | | | |

All primary outcome analyses are adjusted for centre.

<sup>&</sup>lt;sup>1</sup> Participants included in the mITT analysis who adhered to the minimum compliance criteria.

# **Statistical Analysis Plan**

<sup>2</sup> Calculated as the mITT risk difference/proportion adhering to the minimum compliance criteria in the active treatment arm

# Table xx Primary outcome analysis with imputation of missing bleeding assessments

| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) | P value |
|---|---|---|---|---|
| Proportion of participants who die or have bleeding of WHO grade 2 or above from day 1 up to study day 30 - n/N (%) | | | | |
| Hazard ratio (95% CI) | | | | |
| Risk difference (95% CI) | | | | |

Table xx Bleeding between platelet count first ≤30 x 10<sup>9</sup>/L and start of trial treatment – n/N (%)

| | Active<br>arm<br>(n=) | Placebo<br>arm<br>(n=) | Overall<br>(n=) |
|---|---|---|---|
| Number of days between platelet count first ≤30 x 10 <sup>9</sup> /L and start of trial treatment - mean (SD) | | | |
| Number of bleeds between platelet count first ≤30 x 10 <sup>9</sup> /L and start of trial treatment - mean (SD) | | | |
| Number of bleeds of grade 2<br>or above between platelet<br>count first ≤30 x 10 <sup>9</sup> /L and<br>start of trial treatment - mean<br>(SD) | | | |

# 5.10 Figures

- CONSORT diagram
- Median platelet count from consent up to study day 30, by treatment arm
- Overall survival from randomisation to study day 120, by treatment arm
- Highest grade of bleeding a participant experiences, by treatment arm

# 6 Statistical Analysis Plan Amendments

# **Statistical Analysis Plan**

### **Revision History:**

| Version | Author | Date | Reason for revision |
|---|---|---|---|
| 1.1 | EC | 13/03/2020 | <ul> <li>Added summary of numbers of participants who discontinued trial treatment during the period oral treatment was unavailable in the UK.</li> <li>Added footnote to interim analysis.</li> <li>Added minor changes to correct typos suggested by Ian Franklin.</li> <li>Agreed by TMG to include ineligible participants randomised in error in the ITT analysis.</li> </ul> |
| | | | - |

#### 7 References

- 1. MPD998 Statistical Analysis and Reporting
- 2. TREATT bleedgrades v1.2 03\_11\_2017
- 3. Collett D. Modelling survival data in medical research. Florida: Chapman & Hall/CRC, 2003.
- 4. Stanworth SJ, Estcourt LJ, Powter G, Kahan B, Dyer C, Choo L, et al. A no-prophylaxis platelet transfusion strategy for hematologic cancers. N Engl J Med. 2013;368(19):1771-80.
- 5. Van Buuren, S. Multiple imputation of discrete and continuous data by fully conditional specification. *Statistical Methods in Medical Research* 2007; 16: 219–242.

### Appendix 1

#### Table xx Reported SAEs

| Pt ID | Treatment arm | Description | Serious criterion | TREATT Classification |
|---|---|---|---|---|

### Table xx Unexpected adverse reactions

| Pt<br>ID | Treatment arm | Description | TREATT Classification | Causality |
|----------|---------------|-------------|-----------------------|-----------|

### Table xx Thrombotic events

| Pt ID | Pt ID Treatment Type of thrombotic event arm | Serious criterion |
|---|---|---|

# **Statistical Analysis Plan**

### Table xx Veno-occlusive disease

| Pt ID Treatment Bilirubin at d | | Bilirubin at diagnosis | Serious criterion |
|---|---|---|---|
| | arm | | |